CLINICAL TRIAL: NCT05420506
Title: Treatment of Obesity Without Surgical Intervention by Reversible Reduction of the Small Intestinal Absorption Area
Brief Title: Nonsurgical Reversible Obesity Treatment (NROT1)
Acronym: NROT1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1005
Record Dates: First submitted 2022-06-10; First posted 2022-06-15 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Morbid Obesity
Keywords: obesity treatment; non-surgical; small intestine; reversible
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NROT1 (Experimental): Intestinal device placement in subjects and their follow up
  Interventions: Device: NROT1

INTERVENTIONS:
Device: NROT1 — Dental anchored intestinal placement of obesity treatment device with endoscopic intervention

SUMMARY:
The present study relates to apparatus and methods that can be applied using non-invasive techniques for effectively reducing nutrient absorption in the small intestines of obese people.

DETAILED DESCRIPTION:
Obesity is a worldwide health problem which may be further worsened by global Corona virus (COVID-19) pandemic. It may cause social, psychological disorders and chronic diseases such as diabetes and cardiac problems.

Surgical and existing non-surgical (e.g., intragastric balloon placement) procedures are well established procedures to cope with the morbid obesity problem. The principle of using these procedures is based on reducing the surface area available for absorption in the stomach or in small intestine, so that weight loss is gradually accomplished.

Recent bariatric surgery procedures (a more complete description of which can be found for example on the website of the American Society for Bariatric Surgery at http://www.asbs.org) involve alteration of a patient's digestive tract including various reversible and malabsorptive bypass procedures such as jejuno-ileal bypass, gastric bypass and Roux-en-Y gastric bypass, or by irreversible gastric sleeve (restrictive) procedures.

In non-surgical intragastric balloon (IGB) placement procedures, the volume of the space occupying device (balloon) prevents the ingestion of food into the stomach, reducing the desire for food.

Most known complications of IGBs are nausea, vomiting, and discomfort, during and/or shortly after their insertion and removal. Blockage risk of the exit of the stomach (pylori) due to squeezing-pushing action of the stomach is another issue with IGBs.

On April 27, 2020, the U.S. Food and Drug Administration (FDA) released an update on the potential risks of over-inflation (spontaneous hyperinflation), acute pancreatitis, and deaths in patients with some liquid-filled IGBs. Hyperinflation involves the spontaneous filling of IGBs with additional air or liquid while the balloon is in the stomach, this usually requires IGB removal. On the other hand, the mechanism of acute pancreatitis development could be related to pressure from the IGB and distended stomach causing direct injury to the pancreatic parenchyma, compression of the pancreatic duct, and/or indirect pancreatic injury through duodenal obstruction.

All of these critical observations mentioned above show that there is a need for a transorally placed device which can be easily inserted into and removed from the gastrointestinal tract, does not migrate, minimize complications, well tolerated and less costly.

The present study aims to provide a gastrointestinal implant device which includes a solid part for placement into a small intestine so that it reduces absorption of nutrients and particularly fats through the small intestine. This can be more effective weight losing procedure than IGB application alone in stomach, as nutrients and fat intake can be reduced using intestinal implant device.

Transorally placed implant device can be easily inserted into and removed from the gastrointestinal tract, does not migrate, and costs less.

While existing non-surgical weight losing devices induce satiation, hence reduce the frequency and amount of eating, present invention does not limit them, since the operational principle of the present study is neither based on a space occupying type nor a sleeve type implant.

SCIENTIFIC BACKGROUND

1. All orally ingested foods with caloric value are absorbed from the small intestine, and especially from the proximal small intestine, then pass into the blood. Colon provides only the absorption of fluid and electrolytes.
2. As the length of the small intestine is shortened, the intestinal absorption area for the foods with caloric value will decrease, so even if the patient continues to eat, he or she does not gain weight, on the contrary, he or she loses weight.
3. When the orally ingested foods pass through the stomach and duodenum and then enter into the small intestine, they are pushed from proximal to distal intestine by segmental contraction and relaxation movements called peristaltic movements. During these movements, if the food remains stable or stuck in a certain intestinal region, the small intestine segments gather into the proximal region of the intestine and try to push the food to distal end of small intestine by making more severe peristaltic movements. Meanwhile, the length of the small intestine shortens, hence the overall small intestinal absorption area decreases.

Based on this fundamental physiological information, in this study, implant piece placed into the small intestine is anchored either in the stomach or in the oral cavity (dental anchoring) with a biocompatible thread, and the small intestine segments are accumulated in the proximal end of the small intestine in the manner of an accordion in the region where implant device is floating, hence shortening its length and reducing the overall small intestinal absorption area.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of morbid obesity
2. Age limits: 18-65 years
3. No history of gastrointestinal surgery
4. Agreement for voluntary participation in the study

Exclusion Criteria:

1. Presence of obesity that is not at the morbid level
2. Those who do not accept to participate in the study
3. Those who have an obstacle to endoscopic intervention
4. Presence of a history of gastrointestinal surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Change of weight in subjects after 6 Months of intestinal device placement | 6 months
  The weight of each subject will be measured and recorded at the time of intestinal device placement and after 6 months of the placement. Then, statistical analysis will be carried out.

CONTACTS AND LOCATIONS:
Overall Officials: Erhan Aysan, M.D., Principal Investigator — Yeditepe University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ng M, Fleming T, Robinson M, Thomson B, Graetz N, Margono C, Mullany EC, Biryukov S, Abbafati C, Abera SF, Abraham JP, Abu-Rmeileh NM, Achoki T, AlBuhairan FS, Alemu ZA, Alfonso R, Ali MK, Ali R, Guzman NA, Ammar W, Anwari P, Banerjee A, Barquera S, Basu S, Bennett DA, Bhutta Z, Blore J, Cabral N, Nonato IC, Chang JC, Chowdhury R, Courville KJ, Criqui MH, Cundiff DK, Dabhadkar KC, Dandona L, Davis A, Dayama A, Dharmaratne SD, Ding EL, Durrani AM, Esteghamati A, Farzadfar F, Fay DF, Feigin VL, Flaxman A, Forouzanfar MH, Goto A, Green MA, Gupta R, Hafezi-Nejad N, Hankey GJ, Harewood HC, Havmoeller R, Hay S, Hernandez L, Husseini A, Idrisov BT, Ikeda N, Islami F, Jahangir E, Jassal SK, Jee SH, Jeffreys M, Jonas JB, Kabagambe EK, Khalifa SE, Kengne AP, Khader YS, Khang YH, Kim D, Kimokoti RW, Kinge JM, Kokubo Y, Kosen S, Kwan G, Lai T, Leinsalu M, Li Y, Liang X, Liu S, Logroscino G, Lotufo PA, Lu Y, Ma J, Mainoo NK, Mensah GA, Merriman TR, Mokdad AH, Moschandreas J, Naghavi M, Naheed A, Nand D, Narayan KM, Nelson EL, Neuhouser ML, Nisar MI, Ohkubo T, Oti SO, Pedroza A, Prabhakaran D, Roy N, Sampson U, Seo H, Sepanlou SG, Shibuya K, Shiri R, Shiue I, Singh GM, Singh JA, Skirbekk V, Stapelberg NJ, Sturua L, Sykes BL, Tobias M, Tran BX, Trasande L, Toyoshima H, van de Vijver S, Vasankari TJ, Veerman JL, Velasquez-Melendez G, Vlassov VV, Vollset SE, Vos T, Wang C, Wang X, Weiderpass E, Werdecker A, Wright JL, Yang YC, Yatsuya H, Yoon J, Yoon SJ, Zhao Y, Zhou M, Zhu S, Lopez AD, Murray CJ, Gakidou E. Global, regional, and national prevalence of overweight and obesity in children and adults during 1980-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2014 Aug 30;384(9945):766-81. doi: 10.1016/S0140-6736(14)60460-8. Epub 2014 May 29. PMID 24880830
- [Background] Daniel S, Soleymani T, Garvey WT. A complications-based clinical staging of obesity to guide treatment modality and intensity. Curr Opin Endocrinol Diabetes Obes. 2013 Oct;20(5):377-88. doi: 10.1097/01.med.0000433067.01671.f5. PMID 23974764
- [Background] Nguyen NT, Vu S, Kim E, Bodunova N, Phelan MJ. Trends in utilization of bariatric surgery, 2009-2012. Surg Endosc. 2016 Jul;30(7):2723-7. doi: 10.1007/s00464-015-4535-9. Epub 2015 Dec 10. PMID 26659240
- [Background] Vargas EJ, Rizk M, Bazerbachi F, Abu Dayyeh BK. Medical Devices for Obesity Treatment: Endoscopic Bariatric Therapies. Med Clin North Am. 2018 Jan;102(1):149-163. doi: 10.1016/j.mcna.2017.08.013. PMID 29156183
- [Background] Sullivan S, Edmundowicz SA, Thompson CC. Endoscopic Bariatric and Metabolic Therapies: New and Emerging Technologies. Gastroenterology. 2017 May;152(7):1791-1801. doi: 10.1053/j.gastro.2017.01.044. Epub 2017 Feb 10. PMID 28192103
- [Background] Nieben OG, Harboe H. Intragastric balloon as an artificial bezoar for treatment of obesity. Lancet. 1982 Jan 23;1(8265):198-9. doi: 10.1016/s0140-6736(82)90762-0. PMID 6119560
- [Background] Stimac D, Klobucar Majanovic S, Belancic A. Endoscopic Treatment of Obesity: From Past to Future. Dig Dis. 2020 Jan 6:1-13. doi: 10.1159/000505394. Online ahead of print. PMID 31905356
- [Background] Kral J, Machytka E, Horka V, Selucka J, Dolecek F, Spicak J, Kovarova V, Haluzik M, Buzga M. Endoscopic Treatment of Obesity and Nutritional Aspects of Bariatric Endoscopy. Nutrients. 2021 Nov 26;13(12):4268. doi: 10.3390/nu13124268. PMID 34959819
- [Background] Chiang AL, Ryou M. Endoscopic treatment of obesity. Curr Opin Gastroenterol. 2016 Nov;32(6):487-491. doi: 10.1097/MOG.0000000000000307. PMID 27607342
- [Background] Swidnicka-Siergiejko A, Wroblewski E, Andrzej D. Endoscopic treatment of obesity. Can J Gastroenterol. 2011 Nov;25(11):627-33. doi: 10.1155/2011/174163. PMID 22059171
- [Background] Familiari P, Boskoski I, Marchese M, Perri V, Costamagna G. Endoscopic treatment of obesity. Expert Rev Gastroenterol Hepatol. 2011 Dec;5(6):689-701. doi: 10.1586/egh.11.77. PMID 22017697
- [Background] Lee HL. Role of Restrictive Endoscopic Procedures in Obesity Treatment. Clin Endosc. 2017 Jan;50(1):17-20. doi: 10.5946/ce.2017.022. Epub 2017 Jan 30. PMID 28147476
- [Background] Park JM. Role of Malabsorptive Endoscopic Procedures in Obesity Treatment. Clin Endosc. 2017 Jan;50(1):26-30. doi: 10.5946/ce.2017.004. Epub 2017 Jan 30. PMID 28147470
- [Background] Hurt RT, Frazier TH, Mundi MS. Novel Nonsurgical Endoscopic Approaches for the Treatment of Obesity. Nutr Clin Pract. 2017 Aug;32(4):493-501. doi: 10.1177/0884533617714235. Epub 2017 Jun 16. PMID 28622478
- [Background] Espinet-Coll E, Nebreda-Duran J, Gomez-Valero JA, Munoz-Navas M, Pujol-Gebelli J, Vila-Lolo C, Martinez-Gomez A, Juan-Creix-Comamala A. Current endoscopic techniques in the treatment of obesity. Rev Esp Enferm Dig. 2012 Feb;104(2):72-87. doi: 10.4321/s1130-01082012000200006. PMID 22372801
- [Background] DeLegge MH. Endoscopic approaches for the treatment of obesity: fact or fiction? Nutr Clin Pract. 2011 Oct;26(5):534-8. doi: 10.1177/0884533611419667. PMID 21947636
- [Background] Carrano FM, Peev MP, Saunders JK, Melis M, Tognoni V, Di Lorenzo N. The Role of Minimally Invasive and Endoscopic Technologies in Morbid Obesity Treatment: Review and Critical Appraisal of the Current Clinical Practice. Obes Surg. 2020 Feb;30(2):736-752. doi: 10.1007/s11695-019-04302-8. PMID 31802407
- [Background] Davis M, Kroh M. Novel Endoscopic and Surgical Techniques for Treatment of Morbid Obesity: A Glimpse into the Future. Surg Clin North Am. 2016 Aug;96(4):857-73. doi: 10.1016/j.suc.2016.03.005. PMID 27473806
- [Background] Ibrahim M, Blero D, Deviere J. Endoscopic options for the treatment of obesity. Gastroenterology. 2010 Jun;138(7):2228-32, 2232.e1. doi: 10.1053/j.gastro.2010.04.030. Epub 2010 Apr 21. No abstract available. PMID 20416311
- [Background] Katakwar A, Lakhtakia S, Rao GV. Response to Five-Year Outcomes of Endoscopic Sleeve Gastroplasty for the Treatment of Obesity. Clin Gastroenterol Hepatol. 2021 Dec;19(12):2685. doi: 10.1016/j.cgh.2020.11.046. Epub 2020 Dec 2. No abstract available. PMID 33278576
- [Background] Maydeo A, Patil G, Dalal A, Thakare S, Iyer A, Patil N. An Indian Experience of Endoscopic Treatment of Obesity by Using a Novel Technique of Endoscopic Sleeve Gastroplasty (Accordion Procedure). J Assoc Physicians India. 2020 Aug;68(8):14-17. PMID 32738834
- [Background] Lopez-Nava G, Galvao MP, Bautista-Castano I, Fernandez-Corbelle JP, Trell M, Lopez N. ENDOSCOPIC SLEEVE GASTROPLASTY FOR OBESITY TREATMENT: TWO YEARS OF EXPERIENCE. Arq Bras Cir Dig. 2017 Jan-Mar;30(1):18-20. doi: 10.1590/0102-6720201700010006. PMID 28489162
- [Background] Singh S, de Moura DTH, Khan A, Bilal M, Chowdhry M, Ryan MB, Bazarbashi AN, Thompson CC. Intragastric Balloon Versus Endoscopic Sleeve Gastroplasty for the Treatment of Obesity: a Systematic Review and Meta-analysis. Obes Surg. 2020 Aug;30(8):3010-3029. doi: 10.1007/s11695-020-04644-8. PMID 32399847
- [Background] Velotti N, Bianco P, Bocchetti A, Milone M, Manzolillo D, Maietta P, Amato M, Buonomo O, Petrella G, Musella M. Acute complications following endoscopic intragastric balloon insertion for treatment of morbid obesity in elderly patients. A single center experience. Minerva Chir. 2020 Apr;75(2):72-76. doi: 10.23736/S0026-4733.18.07712-X. Epub 2018 Apr 13. PMID 29658677
- [Background] Verlaan T, de Jong K, de la Mar-Ploem ED, Veldhuyzen EA, Mathus-Vliegen EM, Fockens P. Trans-oral Endoscopic Restrictive Implant System: endoscopic treatment of obesity? Surg Obes Relat Dis. 2016 Nov;12(9):1711-1718. doi: 10.1016/j.soard.2016.02.027. Epub 2016 Mar 2. PMID 27317594
- [Background] Zurawinski W, Sokolowski D, Krupa-Kotara K, Czech E, Sosada K. Evaluation of the results of treatment of morbid obesity by the endoscopic intragastric balloon implantation method. Wideochir Inne Tech Maloinwazyjne. 2017;12(1):37-48. doi: 10.5114/wiitm.2017.66856. Epub 2017 Mar 30. PMID 28446931
- [Background] Glass J, Chaudhry A, Zeeshan MS, Ramzan Z. New Era: Endoscopic treatment options in obesity-a paradigm shift. World J Gastroenterol. 2019 Aug 28;25(32):4567-4579. doi: 10.3748/wjg.v25.i32.4567. PMID 31528087
- [Background] Kim SH, Chun HJ. Endoscopic Treatment for Obesity: New Emerging Technology Trends. Gut Liver. 2015 Jul;9(4):431-2. doi: 10.5009/gnl15125. No abstract available. PMID 26087857